CLINICAL TRIAL: NCT02382549
Title: A TRIAL TO EVALUATE THE SAFETY AND IMMUNOGENICITY OF A HELPER PEPTIDE VACCINE PLUS COMBINATION OF BRAF INHIBITION AND MEK INHIBITION (MEL61)
Brief Title: A Clinical Trial to Evaluate a Melanoma Helper Peptide Vaccine Plus Dabrafenib and Trametinib
Acronym: Mel61
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: The study was terminated because of slow accruals.
Sponsor: Craig L Slingluff, Jr (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Craig L Slingluff, Jr, Professor of Surgery and Director, Human Immune Therapy Center, University of Virginia
Organization: University of Virginia (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17700; R01CA178846 (NIH)
Record Dates: First submitted 2015-03-02; First posted 2015-03-06 (Estimated); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Melanoma
Keywords: vaccine; peptide; dabrafenib; trametinib; Montanide ISA-51; MEKINIST; Tafinlar; BRAF inhibitor; MEK inhibitor; BRAFi; MEKi; encorafenib; binimetinib; BRAFTOVI; MEKTOVI; vemurafenib; Zeldoraf; cobimetinib; Cotellic; 6MHP
MeSH Terms: conditions — Melanoma | interventions — MEK inhibitor I

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 6MHP and MEKi and BRAFi (Experimental): The vaccine drug product, 6MHP, consists of 6 class II MHC-restricted peptides derived from melanoma proteins. Each vaccine consists of 200 mcg of each of the six peptides. An aqueous solution of vaccine is mixed 1/1 with Montanide ISA-51 to form water-in-oil emulsions. Vaccines are administered days 1, 8, 15, 36, 57, 78. All peptide vaccines are administered intradermally and subcutaneously.
  A selective BRAF inhibitor and a selective MEK inhibitor will be administered in accordance with the prescribing information.
  Interventions: Drug: BRAF inhibitor; Biological: 6MHP; Drug: MEK inhibitor

INTERVENTIONS:
Drug: BRAF inhibitor — BRAF inhibitor
Biological: 6MHP — 6 melanoma helper vaccine comprised of 6 class II MHC-restricted helper peptides
  Other Names: 6 melanoma helper peptide vaccine
Drug: MEK inhibitor — MEK Inhibitor

SUMMARY:
This study evaluates whether it is safe to administer a helper peptide vaccine with BRAF inhibitor and MEK inhibitor therapy. This study will also evaluate the effects of the combination of the peptide vaccine and BRAF inhibitors/MEK inhibitors on the immune system. We will monitor these effects by performing tests in the laboratory on participants' blood and tumor samples.

ELIGIBILITY:
Inclusion Criteria:

Cohort 1 (Advanced): Measurable stage IIIB, IIIC, IIID or IV melanoma with clinical or radiological evidence of disease. These participants may have had cutaneous, uveal, mucosal primary melanoma, or an unknown primary melanoma. Staging must be confirmed by cytological or histological examination. Staging of cutaneous melanoma will be based on the revised AJCC 8th Edition staging system (Appendix 2) 66.

Cohort 2 (Neo-adjuvant): Resectable stage IIIB, IIIC, IIID, or IV melanoma at initial presentation or subsequent recurrence. These participants have disease amenable to complete surgical resection at the time of enrollment in the study. The resectable disease does not need to be measurable by RECIST v1.1 criteria.

Cohort 3 (Adjuvant): Participants with stage IIIA, IIIB, IIIC, IIID or IV melanoma resected to no evidence of disease. Participants must initiate therapy within 12 weeks of last surgical resection and within 12 weeks of being rendered clinically free of disease by non-surgical approaches Patients that have undergone ablative therapy to a metastatic lesion (e.g. GKRS, radiofrequency ablation) that manifest no additional sites of disease at enrollment are eligible for treatment on cohort 3

* Participants must be eligible to be treated with BRAF inhibitor and MEK inhibitor combination.
* Participants with prior therapy with targeted therapies specific for mutated BRAF including BRAF and/or MEK inhibitors are eligible provided that there was clinical benefit to prior therapy with these agents as judged by the treating physician. There must be an interval of at least 6 months from the last BRAF/MEK therapy and enrollment in this clinical study
* Participants will be required to have radiological studies at baseline to establish measurable disease for cohort 1 or to prove lack of distant metastases for cohorts 2 and 3. Required studies include:

  * Chest CT scan,
  * Abdominal and pelvic CT scan, and
  * Head CT scan or MRI
* Participants in cohorst 1 & 2 who have metastatic melanoma safely available for biopsy pretreatment and on day 22 must consent to having those biopsies. These metastases may be in nodes, skin, soft tissue, liver, or other sites that can be accessed by needle biopsy, incisional or excisional biopsy, with or without image guidance.
* 3.1.6 Participants who have had brain metastases will be eligible if all of the following are true:

  * Each brain metastasis must have been completely removed by surgery or each unresected brain metastasis must have been treated with stereotactic radiosurgery or systemic immunotherapy
  * There has been no evident growth of any brain metastasis since the most recent treatment if the last treatment is >4 weeks prior to enrollment
  * No brain metastasis is > 2 cm in diameter at the time of registration
  * Neurologic symptoms have returned to baseline off steroids,
  * Subjects are not using steroids for at least 7 days prior to registration.
  * The most recent surgical resections or gamma-knife therapy for malignant melanoma must have been completed ≥ 1 week prior to registration
* ECOG performance status of 0-2
* Participants must have the ability and willingness to give informed consent
* Laboratory parameters as follows:

  * ANC > 1000/mm3
  * Platelets > 100,000/mm3
  * Hgb > 9 g/dL
  * HgB-A1c ≤ 8.5%
  * AST and ALT up to 2.5 x upper limits of normal (ULN). Patients known to have Gilbert's disease may be eligible with AST and ALT up to 5 x ULN.
  * Bilirubin up to 2.5 x ULN
  * Alkaline phosphatase up to 2.5 x ULN.
  * Creatinine up to 1.5 x ULN
* Age 18 years or older at registration
* Participants must have at least two intact (undissected) axillary and/or inguinal lymph node basins

Exclusion Criteria:

* Participants who have received the following medications or treatments at any time within 4 weeks of registration:

  * • Chemotherapy
  * Interferon (e.g. Intron-A®)
  * Radiation therapy (Stereotactic radiotherapy, such as gamma knife, can be used ≥ 1 week and ≤ 6 months prior to registration)
  * Allergy desensitization injections
  * Corticosteroids, administered transdermally, parenterally or orally. Inhaled steroids (e.g.: Advair®, Flovent®, Azmacort®) are not permitted. Topical corticosteroids are acceptable.
  * Growth factors (e.g. Procrit®, Aranesp®, Neulasta®)
  * Interleukins (e.g. Proleukin®)
  * Any investigational medication
* HIV positivity or evidence of active Hepatitis C virus.
* Participants who are currently receiving nitrosoureas or who have received this therapy 6 weeks prior to registration
* Participants who are currently receiving a checkpoint molecule blockade therapy, or who have received this therapy within 3weeks prior to registration.
* Participants with known or suspected allergies to any component of the vaccine.
* Participants may not have been vaccinated previously with any of the synthetic peptides included in this protocol. Participants who have received vaccinations containing agents other than the synthetic peptides included in this protocol and have recurred during or after administration of the vaccine will be eligible to enroll 12 weeks following their last vaccination.
* Pregnancy.
* Female participants must not be breastfeeding
* Participants in whom there is a medical contraindication or potential problem in complying with the requirements of the protocol in the opinion of the investigator.
* Participants classified according to the New York Heart Association classification as having Class III or IV heart disease.
* Participants with uncontrolled diabetes, defined as having a HgB-A1c greater than 7.5%.
* Participants must not have had prior autoimmune disorders requiring cytotoxic or immunosuppressive therapy, or autoimmune disorders with visceral involvement. Participants with an active autoimmune disorder requiring these therapies are also excluded.
* Participants who have another cancer diagnosis, except that the following diagnoses will be allowed:

  * squamous cell cancer of the skin without known metastasis
  * basal cell cancer of the skin without known metastasis
  * carcinoma in situ of the breast (DCIS or LCIS)
  * carcinoma in situ of the cervix
  * any cancer without distant metastasis that has been treated successfully, without evidence of recurrence or metastasis for over 3 years
* Participants with known addiction to alcohol or drugs who are actively taking those agents, or participants with recent (within 1 year of registration) or ongoing illicit IV drug use.
* Body weight < 110 pounds
* Participants with a known history of glucose-6-phosphate dehydrogenase deficiency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-04; Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Adverse event profile for the combination of BRAFi, MEKi, and 6MHP | 30 days after the last vaccination with 6MHP
CD4+ T cell responses in the blood | through day 85
  CD4+ T cell responses to the peptide vaccine

SECONDARY OUTCOMES:
An evaluation of the infiltration of T cells into melanoma metastases pre and post-vaccination. | pre-vaccine and day 22
Antibody responses against 6MHP | through day 85
  An evaluation of the development of antibdoy responses following vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Gaughan, MD, Principal Investigator — University of Virginia; Craig L. Slingluff, Jr., MD, Study Director — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States